CLINICAL TRIAL: NCT03972748
Title: Evaluation Of The Treatment With Oral Itraconazole In Patients With Basocellular Carcinoma Of Skin, Locally Limited Disease.
Brief Title: Use Of Oral Itraconazole In Patients With Locally Limited Basocellular Carcinoma Of Skin.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47011715.0.0000.5327
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Basal Cell Carcinoma; Hedgehog Pathway
Keywords: Itraconazole
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Itraconazole (Experimental): Oral Itraconazole capsules, 200 mg
  Interventions: Drug: Itraconazole 200 mg

INTERVENTIONS:
Drug: Itraconazole 200 mg — Oral Itraconazole capsules, 200 mg, twice daily, for 60 days prior to surgery with curative intent.

SUMMARY:
Patients with localized basocellular carcinoma of the skin, will receive oral Itraconazole, 200 mg twice daily, for 60 days, prior to curative intent surgery.

DETAILED DESCRIPTION:
Patients with localized basocellular carcinoma of the skin, will receive oral Itraconazole, 200 mg once daily, for 60 days, before surgery with curative intent.

Tumor area regression will be measured through dermatologic evaluation and photographic documentation on baseline and at the end of the 60 day treatment period.

The activity of the Hedgehog pathway will be measured on tissue samples obtained at the time of diagnosis and at the time of curative intent surgery, through the measuring of the Ki67 index.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of Basocellular Carcinoma (BCC) of the Skin, histologically confirmed.
* At least one BCC lesion with 10 mm in the longest diameter
* Disease amenable to surgical intervention with curable intent.
* Signed Informed Consent
* PS ECOG 0 to 3

Exclusion Criteria:

* Chronic renal disease, with a glomerular filtration rate of less than 30 ml/min
* Acute or chronic liver disease, as measured by: total bilirubin > than 1.5 x ULN and AST and ALT > than 5 x ULN.
* Symptomatic cardiac insufficiency or an ejection fraction lower than 50% measured through echocardiography,
* Other active malignancies in the last year.
* Uncontrolled systemic hypertension,
* Any chronic infections such as tuberculosis, viral hepatitis and HIV.
* Pregnancy, suspected or confirmed.
* Known intolerance to the use of Itraconazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
clinical response | 60 days
  tumor area response registered through dermatologic evaluation
hedgehog pathway activity | 60 days
  Measured through the Ki67 index on pathological specimens at the beginning and at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Renato M Bakos, Ph. D., Study Chair — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided